CLINICAL TRIAL: NCT06855290
Title: Tumor Immunity and Cancer Recurrence Prediction Model
Status: Not yet recruiting | Type: Observational
Sponsor: Anhui Provincial Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: KY2021204
Record Dates: First submitted 2025-02-23; First posted 2025-03-03 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Cancer
Keywords: cancer; immunity; tumor
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Surgical resection of tumor tissue samples (The tumor tissue will not be used for DNA extraction).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The purpose of this observational study is to understand the predictive effect of the laboratory-developed TIMES scoring system on the recurrence status of cancer patients who have undergone surgical tumor resection. The main questions it aims to answer are:

Can the TIMES scoring system accurately predict the recurrence status of cancer patients who have undergone surgical tumor resection? What is the accuracy of the TIMES scoring system? The medical records or biological specimens used in this study were obtained from previous clinical treatments, and the tissues used were collected from post-surgical discarded tissues from the participants, which will not affect their health. Researchers will continuously monitor the disease progression of the participants for up to 10 years or until cancer recurrence occurs.

DETAILED DESCRIPTION:
No grouping, the long-term tracking of participants' disease progression and recurrence status will be compared with the analysis results of the collected discarded tumor tissues from the participants' surgeries

ELIGIBILITY:
Inclusion Criteria：

1.Adult males and females (non-pregnant, non-lactating)； 2.18 years or older (inclusive); 3.Diagnosis: Diagnosed with cancer (e.g., liver cancer, lung cancer, gastric cancer, colorectal cancer, etc.) and eligible for surgical resection; 4.Informed Consent: Participants must be fully informed about the study prior to participation and voluntarily sign a written informed consent form;

Exclusion Criteria：

1. Specimens from pregnant or lactating patients will not be included in this study, and participant should have no plans for pregnancy or lactation within the next 2 years.
2. Participants must be at least 18 years old.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants must be at least 18 years old, not pregnant, and not breastfeeding, diagnosed with cancer (such as liver cancer, lung cancer, gastric cancer, colorectal cancer, etc.), and eligible for surgical resection
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
recurrence | From the date of random grouping to the date of first recorded recurrence or death due to any reason, whichever comes first, the evaluation lasts up to 120 months.
  The time from when the participant undergoes surgical treatment to the recurrence of cancer, which is obtained by researchers through phone follow-ups.
disease-free progression period | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 120 months
  The time from when the participant undergoes surgical treatment to any progression of cancer, which is obtained by researchers through phone follow-ups.
RECIST1.1 | From the start of clinical treatment to the end of clinical treatment, up to a maximum of 120 months.
  Tumor size: Measure the longest diameter or maximum cross-sectional area of the target tumor and record its changes.
  Evaluation criteria:
  Complete Response (CR): All target lesions disappear. Partial Response (PR): The tumor's maximum diameter or volume decreases by at least 30%.
  Stable Disease (SD): The tumor shows no significant growth or shrinkage, with changes within a certain range.
  Progressive Disease (PD): The tumor's maximum diameter or volume increases by at least 20%.